CLINICAL TRIAL: NCT06797622
Title: An Open-label Positron Emission Tomography (PET) Study to Investigate the Heterogeneity of 68Ga-FAPI Uptake Predicting the Response of T-DXd Treatment for Brain Metastasis in Patients with HER2-positive Advanced or Metastatic Breast Cancer.
Brief Title: Heterogeneity of 68Ga-FAPI Uptake As Imaging Biomarker in T-DXd Treatment for Brain Metastasis of HER2 Positive Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YOUNGBC-33
Record Dates: First submitted 2025-01-23; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trastuzumab deruxtecan (T-DXd) (Experimental): Trastuzumab deruxtecan (T-DXd)
  Interventions: Drug: Trastuzumab deruxtecan (T-DXd)

INTERVENTIONS:
Drug: Trastuzumab deruxtecan (T-DXd) — Trastuzumab deruxtecan (T-DXd)

SUMMARY:
The purpose of this study was to explore the predictive value of the heterogeneity of 68Ga-FAPI PET-CT uptake before treatment on the response of T-DXd treatment in patients with brain metastases of HER2-positive breast cancer. The patient underwent 68Ga-FAPI PET-CT examinations within 2 weeks before and after 2 cycles of T-DXd treatment. Heterogeneity index, SUVmax, SUVmean and other uptake values were collected to investigate the association with efficacy of T-DXd.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 18 years old.
2. ECOG 0-2.
3. Patients have been diagnosed with unresectable, locally advanced or metastatic HER2-positive breast cancer, which were by means of immunohistochemical analysis (with 3+ indicating positive status), fluorescence in situ hybridization (with an amplification ratio ≥2.0 indicating positive status), or both.
4. Brain metastasis was confirmed by MRI; measurable disease as defined by at least one intracranial cerebral metastatic lesion with diameter ≥ 1.0 cm not previously treated with radiation.
5. It is allowed to use mannitol, bevacizumab, or corticosteroids before enrollment, but dose should be stable for at least one week.
6. Plan to receive Trastuzumab deruxtecan (T-DXd).
7. Adequate bone marrow, liver, kidney and cardiac function.
8. All patients can provide an informed consent before enrolment and data collection.

Exclusion Criteria:

1. Leptomeningeal involvement.
2. Uncontrolled large amount of pleural effusion and ascites.
3. Previous treatment of T-DXd.
4. Adequate treatment washout period before enrollment, defined as: major surgery ≥4 weeks, radiation therapy ≥4 weeks, chemotherapy ≥4 weeks, small-molecule targeted agents, anticancer hormonal therapy, antibody-based treatment ≥3 weeks.
5. Patients with previous interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis require corticosteroids treatment; or any clinically active interstitial lung disease currently.
6. Use of any investigational agent within 14 d before initiation of treatment.
7. Concomitant other anticancer therapy, including cytotoxic, targeted agents, immunotherapy, antibody, retinoid or anticancer hormonal treatment.
8. History of malignancy other than squamous cell carcinoma, basal cell carcinoma of the skin or carcinoma in situ of the cervix within the last 3 years, including contralateral breast cancer.
9. Clinically significant cardiac disease.
10. Patients with known hypersensitivity to trastuzumab or 68Ga-FAPI.
11. a history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to study drugs.
12. Patients with the history of immunodeficiency, including HIV, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
13. Patients with HBsAg positive and HBV >=1000, HCV antibody positive, TP-Ab positive or HIV positive.
14. Pregnant or lactating women. Women with childbearing potential must have a negative pregnancy test at screening; also excluded are women with childbearing potential, including women whose last menstrual period was <1 year before screening, unable or unwilling to use adequate contraception from study start to 1 year after the last dose of protocol therapy. Acceptable contraception methods included the application of an intrauterine device, barrier method or total abstinence.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Difference of baseline heterogeneity index | 6 weeks
  Difference of baseline heterogeneity index evaluated by 68Ga-FAPI PET-CT between cerebral lesions reaching ORR or not with the T-DXd treatment.

SECONDARY OUTCOMES:
68Ga-FAPI PET-CT value | 6 weeks
  68Ga-FAPI PET-CT value changes (SUVmax, SUVmean ) at baseline and 2 cycles after T-DXd treatment of brain metastasis lesions.
Difference of baseline heterogeneity index | 6 weeks
  Difference of baseline heterogeneity index evaluated by 68Ga-FAPI PET-CT for PFS, CBR and OS in patients with brain metastasis after the T-DXd treatment.
Difference of baseline heterogeneity index | 6 weeks
  Difference of baseline heterogeneity index, SUVmax and SUVmean evaluated by 68Ga-FAPI PET-CT between active or stable brain metastasis.
68Ga-FAPI PET-CT value | 6 weeks
  68Ga-FAPI PET-CT value changes (heterogeneity index, SUVmax, SUVmean ) at baseline and 2 cycles after T-DXd treatment of whole body metastasis lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Profssor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China